CLINICAL TRIAL: NCT00095563
Title: A Phase 2 Study of GW572016 in Recurrent and/or Metastatic Adenoid Cystic Carcinoma, and Other EGFR-and/or erbB2-expressing Malignant Tumors of the Salivary Glands
Brief Title: Lapatinib in Treating Patients With Recurrent and/or Metastatic Adenoid Cystic Cancer or Other Salivary Gland Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03089; NCI-2012-03089 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 6701; PHL-028 (Other: Princess Margaret Hospital Phase 2 Consortium); 6701 (Other: CTEP); N01CM62201 (NIH); N01CM62203 (NIH)
Record Dates: First submitted 2004-11-05; First posted 2004-11-08 (Estimated); Results first posted 2017-04-18 (Actual); Last update posted 2017-04-18 (Actual); Status verified 2017-03

CONDITIONS: High-grade Salivary Gland Carcinoma; High-grade Salivary Gland Mucoepidermoid Carcinoma; Low-grade Salivary Gland Carcinoma; Low-grade Salivary Gland Mucoepidermoid Carcinoma; Recurrent Adenoid Cystic Carcinoma of the Oral Cavity; Recurrent Salivary Gland Cancer; Salivary Gland Acinic Cell Tumor; Salivary Gland Adenocarcinoma; Salivary Gland Adenoid Cystic Carcinoma; Salivary Gland Malignant Mixed Cell Type Tumor
MeSH Terms: conditions — Salivary Gland Neoplasms | interventions — Lapatinib; N-(3-chloro-4-((3-fluorobenzyl)oxy)phenyl-6-(5-((methylsulfonyl)ethyl)aminomethyl)-2-furyl)-4-quinazolinamine

ARMS (1):
- Treatment (lapatinib ditosylate) (Experimental): Patients receive oral lapatinib once daily on days 1-28. Courses repeat every 28 days in the absence of unacceptable toxicity or disease progression.
  Interventions: Drug: lapatinib ditosylate; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: lapatinib ditosylate — Given orally
  Other Names: GSK572016; GW-572016; GW2016; Lapatinib; Tykerb
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase II trial to study the effectiveness of lapatinib in treating patients who have recurrent and/or metastatic adenoid cystic cancer or other salivary gland cancers. Lapatinib may stop the growth of tumor cells by blocking the enzymes necessary for their growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the antitumor activity of GW572016 in recurrent and/or metastatic adenoid cystic carcinoma of the salivary glands using objective response rates (partial and complete responses).

SECONDARY OBJECTIVES:

I. To determine the duration of objective response, rate and duration of stable disease, progression-free, median and overall survival rates of GW572016 in recurrent and/or metastatic adenoid cystic carcinoma of the salivary glands.

II. To estimate the antitumor activity of GW572016 in other epidermal growth factor receptor (EGFR)- and/or erbB2-overexpressing malignant tumors of the salivary glands using objective response rates (partial and complete responses).

III. To document the safety and tolerability of GW572016 in these patient populations

TERTIARY OBJECTIVES:

I. To investigate if differences in baseline levels of EGFR and/or erbB2 expression, and receptor phosphorylation status in tumor specimens predict outcome to therapy.

II. To investigate if the inhibitory effects of GW572016 on EGFR and/or erbB2 pathway activation in tumor specimens correlate with clinical outcome.

III. To determine the steady state levels of GW572016 achieved, and their correlation with clinical and laboratory correlative endpoints.

OUTLINE: This is a nonrandomized, open-label, multicenter study.

Patients receive oral lapatinib once daily on days 1-28. Courses repeat every 28 days in the absence of unacceptable toxicity or disease progression.

Patients are followed for survival

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically documented or cytologically confirmed adenoid cystic, or other malignant salivary gland carcinomas of major or minor salivary gland origin; all patients must have either EGFR and/or erbB2 expressing tumors (for definitions of EGFR and erbB2 expression to be enrolled in this study; EGFR and erbB2 expression will be determined using archival paraffin samples for all study patients where possible; if these samples are unavailable then patients must undergo a biopsy to determine their EGFR and erbB2 status
* Patients must have recurrent and/or metastatic disease that is progressive and not amenable to surgery or curative radiotherapy; progressive disease is defined as one of the following occurring within 6 months of study entry:

  * At least a 20% increase in radiologically or clinically measurable disease
  * Appearance of any new lesions or
  * Deterioration in clinical status
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral CT scan
* Patients may have had unlimited prior therapy; however, there must be at least a 4 weeks' interval between any chemotherapy (6 weeks for nitrosoureas or mitomycin C), radiotherapy or surgery and study enrollment; exceptions may be made however, for low dose, non-myelosuppressive radiotherapy - please contact the Principal Investigator (Dr. L. Siu) PRIOR to registration if questions arise about the interpretation of this criterion; for patients who received local therapy prior to study entry, there must be either progression of measurable disease documented within the treatment field, or must have measurable disease outside the treatment field prior to study entry
* Life expectancy of greater than 12 weeks
* ECOG performance status 0,1, or 2
* Leukocytes >= 3,000/uL
* Absolute neutrophil count >= 1,5000/uL
* Platelets >= 100,000/uL
* Total bilirubin within normal institutional limits
* AST(SGOT)/ALT(SGPT) =< 2.5 x institutional upper limit of normal
* Creatinine within normal institutional limits OR
* Creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Cardiac ejection fraction within the institutional range of normal as measured by echocardiogram or MUGA scan: Note that baseline and on treatment scans should be performed using the same modality and preferably at the same institution
* Must be willing and able to undergo tumor biopsy once before and once during investigational therapy; patients must have tumor lesions accessible for biopsy for correlative studies; the decision regarding the safety of doing a biopsy will be made by an interventional radiologist rather than the investigator and must be documented in writing; in cases where there is a medical contraindication to tumor biopsy, exception may be granted only upon discussion with the principal investigator
* Eligibility of patients receiving medications or substances known to affect, or with the potential to affect the activity or pharmacokinetics of GW572016 will be determined following review of their use by the principal investigator; a list of medications and substances known or with the potential to interact with CYP450 isoenzymes is provided in: Cytochrome P-450 Enzymes and Drug metabolism; in: Lacy CF, Armstrong LL, Goldman MP, Lance LL eds; Drug Information Handbook 8TH ed. Hudson, OH; LexiComp Inc. 2000: 1364-1371
* HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with GW572016; appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated
* Patients requiring oral anticoagulants (coumadin, warfarin) are eligible provided there is increased vigilance with respect to monitoring INR; if medically appropriate and treatment available, the investigator may also consider switching these patients to LMW heparin, where an interaction with GW572016 is not expected
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document
* Able to swallow and retain oral medication; alternately, for patients who require feeding via nasogastric tubes or who cannot swallow whole tablets, study entry is allowed by following instructions on drug administration

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or
* Patients who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients who have had prior treatment with EGFR or erbB2 targeting therapies
* Patients may not be receiving any other investigational agents or receiving concurrent anticancer therapy
* Patients with known brain metastases but have remained stable for at least 3 months since completion of radiotherapy or surgery, have no significant neurological deficits, and are off corticosteroids, may be allowed on study; patients with symptomatic brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* Patients with a history of other active malignancy in the past 5 years (with the exception of adequately treated cervical carcinoma in situ and non-melanomatous skin cancers) are excluded
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to GW572016
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because GW572016 is member of the 4-anilinoquinazoline class of kinase inhibitors with the potential for teratogenic or abortifacient effects; breastfeeding should be discontinued if the mother is treated with GW572016
* HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study
* Patients with GI tract disease resulting in an inability to take oral medication, malabsorption syndrome, a requirement for IV alimentation, prior surgical procedures affecting absorption, uncontrolled inflammatory GI disease (e.g., Crohn's, ulcerative colitis)
* Concomitant requirement for medication classified as CYP3A4 inducer or inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2004-09; Primary Completion 2009-02 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Siu, Principal Investigator — Princess Margaret Hospital Phase 2 Consortium
Locations (1):
- Princess Margaret Hospital Phase 2 Consortium, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 enrolled patient was a screen failure.
Period: Overall Study
Arm/Group | Treatment (Lapatinib Ditosylate)
Started | 39
Completed | 39
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Lapatinib Ditosylate)
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 13
Age, Continuous [Median (Full Range); unit: years] | 57 [39 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 29
Region of Enrollment [Number; unit: participants]
  Canada | 40

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rates (Partial and Complete Responses)
Description: Per Response - Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions;
Time Frame: Up to 5 years
Population: 36 assessable participants.
Measure: Number; unit: participants
Arm/Group | Treatment (Lapatinib Ditosylate)
Number analyzed (Participants) | 36
participants | 0

2. Secondary Outcome: Duration of Objective Response
Time Frame: From the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented, assessed up to 5 years
Population: This assessment was not performed since no participants showed a response.
Arm/Group | Treatment (Lapatinib Ditosylate)
Number analyzed (Participants) | 0

3. Secondary Outcome: Rate of Stable Disease
Description: Number of patients who had Stable disease for more than or equal to 6 months together in both Adenoid cystic carcinoma (ACC) and non-adenoid cyctic carcinoma (non-ACC)
Time Frame: 6 months
Population: 36 assessable participants, 19 with ACC and 17 with non-ACC.
Measure: Number; unit: participants
Arm/Group | Treatment (Lapatinib Ditosylate)
Number analyzed (Participants) | 36
participants
  ACC: number analyzed (Participants) | 19
  ACC | 9
  Non-ACC: number analyzed (Participants) | 17
  Non-ACC | 4

4. Secondary Outcome: Progression-free Survival (PFS) According to RECIST
Time Frame: From the date of study enrolment to disease progression, death or last contact, or last tumor assessment before the start of further anti-tumor therapy, assessed up to 5 years
Population: 36 assessable participants, 19 with ACC and 17 with non-ACC.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Lapatinib Ditosylate)
Number analyzed (Participants) | 36
months
  ACC: number analyzed (Participants) | 19
  ACC | 3.6 [3.1 to 12.4]
  Non-ACC: number analyzed (Participants) | 17
  Non-ACC | 2.1 [1.6 to 9.2]

5. Secondary Outcome: Overall Survival (OS)
Description: Survival estimates will be computed using the Kaplan-Meier method.
Time Frame: From the date of study enrolment to death or last contact, assessed up to 5 years
Population: 20 participants with ACC, 19 participants with non-ACC.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Lapatinib Ditosylate)
Number analyzed (Participants) | 39
months
  ACC: number analyzed (Participants) | 20
  ACC | NA [NA to NA] — Not reached
  Non-ACC: number analyzed (Participants) | 19
  Non-ACC | 16.5 [9.1 to 30.9]

6. Secondary Outcome: Most Frequent Adverse Events of Grade 1-2 by CTCAE Grading
Description: Number of participants that experienced the most frequent adverse events of grade 1-2 by CTCAE grading.
Time Frame: Up to 5 years
Measure: Number; unit: participants
Arm/Group | Treatment (Lapatinib Ditosylate)
Number analyzed (Participants) | 39
participants
  Diarrhea | 26
  Fatigue | 28
  Rash | 19

ADVERSE EVENTS:
Arm/Group | Treatment (Lapatinib Ditosylate)
Serious Adverse Events (participants affected / at risk) | 6/39
Other Adverse Events (participants affected / at risk) | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Lapatinib Ditosylate) (N=39)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Hearing loss (Ear and labyrinth disorders) | 1
Ureteric obstruction (Renal and urinary disorders) | 1
Weight gain (Investigations) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Hypertension (Vascular disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Lapatinib Ditosylate) (N=39)
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 4
Activated partial thromboplastin time prolonged (Investigations) | 4
Alanine aminotransferase increased (Investigations) | 8
Alkaline phosphatase increased (Investigations) | 12
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 5
Alopecia (Skin and subcutaneous tissue disorders) | 4
Anorexia (Metabolism and nutrition disorders) | 10
Anxiety (Psychiatric disorders) | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Aspartate aminotransferase increased (Investigations) | 12
Ataxia (Nervous system disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 7
Bilirubin increased (Investigations) | 6
Blood glucose increased (Metabolism and nutrition disorders) | 16
Blood uric acid increased (Metabolism and nutrition disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 4
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Burning in feet (Nervous system disorders) | 1
Cheilitis (Gastrointestinal disorders) | 2
Chest pain (General disorders) | 6
Chest wall pain (General disorders) | 2
Coagulopathy - PT (Investigations) | 1
Constipation (Gastrointestinal disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 14
Creatinine increased (Investigations) | 4
Cyst on back (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Depression (Psychiatric disorders) | 3
Dermatitis radiation (Injury, poisoning and procedural complications) | 1
Diarrhea (Gastrointestinal disorders) | 26
Diplopia (Eye disorders) | 1
Dizziness (Nervous system disorders) | 4
Dry eye syndrome (Eye disorders) | 1
Dry lips (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 12
Dyspepsia (Gastrointestinal disorders) | 11
Dysphagia (Gastrointestinal disorders) | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 18
Dysuria (Renal and urinary disorders) | 2
Ear, nose and throat examination abnormal (General disorders) | 4
Early Satiety (Gastrointestinal disorders) | 1
Edema limbs (General disorders) | 5
Erectile dysfunction (Reproductive system and breast disorders) | 1
External ear inflammation (Ear and labyrinth disorders) | 2
Eye infection (Infections and infestations) | 2
Eye pain (Eye disorders) | 1
Facial nerve disorder (Nervous system disorders) | 1
Facial pain (General disorders) | 3
Fatigue (General disorders) | 28
Fever (General disorders) | 2
Flu-like symptoms (General disorders) | 1
Flushing (Vascular disorders) | 1
Folliculitis (Skin and subcutaneous tissue disorders) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Headache (Nervous system disorders) | 10
Hearing loss (Ear and labyrinth disorders) | 4
Hemoglobin decreased (Investigations) | 20
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 5
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2
INR increased (Investigations) | 1
Insomnia (Psychiatric disorders) | 11
Joint pain (Musculoskeletal and connective tissue disorders) | 3
Kidney infection (Infections and infestations) | 1
Knee injury (Injury, poisoning and procedural complications) | 1
Laryngitis (Respiratory, thoracic and mediastinal disorders) | 1
Left Ear Drainage (Infections and infestations) | 1
Left ventricular failure (Cardiac disorders) | 1
Leukocyte count decreased (Blood and lymphatic system disorders) | 11
Localized edema (General disorders) | 1
Loss Of Peripheral Vision (Eye disorders) | 1
Lymphocyte count decreased (Investigations) | 25
Menopausal symptoms (Reproductive system and breast disorders) | 1
Mucosal infection (Infections and infestations) | 1
Mucositis oral (Gastrointestinal disorders) | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Nail disorder (Skin and subcutaneous tissue disorders) | 3
Nail infection (Infections and infestations) | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4
Nausea (Gastrointestinal disorders) | 16
Neck pain (Musculoskeletal and connective tissue disorders) | 5
Neck soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1
Neuralgia (Nervous system disorders) | 2
Neutrophil count decreased (Investigations) | 7
Nystagmus (Nervous system disorders) | 1
Onycolysis (Skin and subcutaneous tissue disorders) | 1
Optic nerve disorder (Nervous system disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Otitis externa (Ear and labyrinth disorders) | 1
Pain (Infections and infestations) | 1
Pain - hands (Musculoskeletal and connective tissue disorders) | 1
Pain - hip (Musculoskeletal and connective tissue disorders) | 2
Pain - jaw (Musculoskeletal and connective tissue disorders) | 1
Pain - left jaw (Musculoskeletal and connective tissue disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 12
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Plantar Wart (Infections and infestations) | 1
Platelet count decreased (Investigations) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 7
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Pyramidal tract syndrome (Nervous system disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 19
Rash desquamating (Skin and subcutaneous tissue disorders) | 5
Salivation (Gastrointestinal disorders) | 1
Second Malignancy, Supraglottic Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Serum albumin decreased (Metabolism and nutrition disorders) | 3
Serum calcium decreased (Metabolism and nutrition disorders) | 3
Serum calcium increased (Metabolism and nutrition disorders) | 5
Serum cholesterol increased (Investigations) | 2
Serum glucose decreased (Metabolism and nutrition disorders) | 1
Serum magnesium decreased (Metabolism and nutrition disorders) | 2
Serum phosphate decreased (Metabolism and nutrition disorders) | 7
Serum potassium decreased (Metabolism and nutrition disorders) | 5
Serum potassium increased (Metabolism and nutrition disorders) | 1
Serum sodium decreased (Metabolism and nutrition disorders) | 5
Serum sodium increased (Metabolism and nutrition disorders) | 2
Sinus bradycardia (Cardiac disorders) | 2
Sinus tachycardia (Cardiac disorders) | 1
Sinusitis (Infections and infestations) | 1
Skin change (Skin and subcutaneous tissue disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 1
Skin-Carbuncle (Skin and subcutaneous tissue disorders) | 1
Speech disorder (Nervous system disorders) | 1
Taste alteration (Nervous system disorders) | 6
Thermal burn (Injury, poisoning and procedural complications) | 1
Thinner Skin Finger Tips (Skin and subcutaneous tissue disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Tooth infection (Infections and infestations) | 1
Toothache (Gastrointestinal disorders) | 2
Tremor (Nervous system disorders) | 2
Trigeminal nerve disorder (Nervous system disorders) | 1
Trismus (Musculoskeletal and connective tissue disorders) | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ulceration - medical intervention not indicated (Gastrointestinal disorders) | 1
Upper aerodigestive tract infection (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 3
Ureteric obstruction (Renal and urinary disorders) | 1
Urinary frequency (Renal and urinary disorders) | 3
Urinary incontinence (Renal and urinary disorders) | 1
Urinary tract infection (Renal and urinary disorders) | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1
Vaginal discharge (Reproductive system and breast disorders) | 1
Vaginal dryness (Reproductive system and breast disorders) | 1
Vaginal hemorrhage (Reproductive system and breast disorders) | 1
Vision blurred (Eye disorders) | 2
Vision Changes (Eye disorders) | 1
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 6
Watering eyes (Eye disorders) | 1
Weight gain (Investigations) | 1
Weight loss (Investigations) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less